CLINICAL TRIAL: NCT07207018
Title: Early Intervention After Traumatic Exposure in Children and Adolescents: a Randomized Controlled Trial of the Effectiveness of Child and Family Traumatic Stress Intervention (CFTSI).
Brief Title: Early Intervention After Traumatic Exposure in Children and Adolescents
Acronym: ADAPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Toulouse (Other); Centre Hospitalier Universitaire de Nīmes (Other); University Hospital, Thuir (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL24_0351
Record Dates: First submitted 2025-02-05; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
Keywords: CFTSI; Adolescents; Children; Post-Traumatic Stress Disorder; Traumatic event
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The study will be multicenter, prospective, controlled, and open-label, with two parallel arms and blinded assessment of the outcome measures. Recruitment will take place among parents consulting for their children at one of the four branches of the Regional Center for Psychotrauma Occitanie (CRPOcc) within three months of the child's exposure to a traumatic event (TE).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CFTSI group (Experimental): CFTSI, a 5-session intervention of 1.5 hours each, with one session per week, will be implemented in the experimental group by psychotherapists trained in CFTSI. CFTSI is a brief, structured, and standardized intervention that includes an initial session with the parents alone, a second session with the child alone, and three family sessions. Additionally, 1 to 3 extra sessions may be conducted as needed to clarify certain points or review specific strategies in detail). There is a detailed CFTSI manual describing the progression of each session and precise questionnaires used in each session to measure the intensity and frequency of symptoms, as well as their progression over time.
  Interventions: Behavioral: CFTSI (Child and Family Traumatic Stress Intervention)
- Control group (Active Comparator): The control group will undergo five sessions of 1.5 hours each, with one weekly session, of non-specific psychological support therapy, focused on the child rather than the family, and aimed at supporting the child and strengthening their daily adaptation. This support therapy is already integrated into the standard practice of the CRPOCC, but will be conducted by psychotherapists from the Montpellier University Hospital who are not trained in CFTSI, to ensure a consistent format that facilitates comparisons between the two groups. The number of sessions may be increased to a total of eight sessions if the clinician determines that additional aspects need to be addressed during the sessions.
  Interventions: Behavioral: non-specific psychological support therapy

INTERVENTIONS:
Behavioral: CFTSI (Child and Family Traumatic Stress Intervention) — CFTSI is a family-centered intervention lasting five to eight sessions, aiming to strengthen parental support for the child by facilitating the identification of the child's typical responses to traumatics events, improving communication between the child and the parent, and teaching coping strategies and behavioral interventions to both parents and children to reduce acute post-traumatic reactions.
  Arms: CFTSI group
Behavioral: non-specific psychological support therapy — non-specific psychological support therapy, focused on the child rather than the family, and aimed at supporting the child and strengthening their daily adaptation. This support therapy is already integrated into the standard practice of the CRPOCC, but will be conducted by psychotherapists from the Montpellier University Hospital who are not trained in CFTSI, to ensure a consistent format that facilitates comparisons between the two groups. The number of sessions may be increased to a total of eight sessions if the clinician determines that additional aspects need to be addressed during the sessions.
  Arms: Control group

SUMMARY:
The aim of this interventional research is to evaluate the effectiveness of CFTSI in reducing post-traumatic symptoms measured using the CPC, child version, at the end of CFTSI treatment in children and adolescents aged between 7 and 17 years, exposed to an ET in the last 3 months. The main question(s) it aims to answer [is/are]:

* CFTSI reduces posttraumatic Child Posttraumatic Stress Checklist (CPC) scores in children exposed to ET, both immediatly after completion of the CFTSI and at 3 months after completion.
* CFTSI reduces post-traumatic scores in parents on the PTSD Checklist for DSM5 (PCL), both immediatly after completion of the CFTSI and at 3 months after completion.
* researchers will compare the reduction in post-traumatic symptoms between participants receiving CFTSI and those receiving non-specific child-centred psychological support. Symptoms will be assessed using the PCL in parents and the CPC in children and adolescents, immediately after completion of the program and again at 3 months after completion.

The participants will be randomised into two groups, one that will undergo CFTSI and one that will undergo supportive psychological therapy. Each participant will receive one session per week over five weeks, and possibly 1 to 3 additional sessions if necessary over a further three weeks, and will then be reviewed three months later.

DETAILED DESCRIPTION:
Individuals and populations worldwide are exposed to extremely high rates of maltreatment, violence, sexual and physical abuse, bullying, severe accidents, and exposure to other traumatic events (TE) such as natural disasters, terrorist attacks, war, and forced migration. The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) defines a traumatic event as any situation involving "actual or threatened death, serious injury, or sexual violence". A report based on epidemiological data from 24 different countries found that 70% of the populations studied worldwide report exposure to at least one TE in their lifetime. This exposure is more frequently observed among children, adolescents, and young adults, with 60% of youth under 18 having experienced at least one TE in the past year.

Childhood traumatic exposure is associated with an increased risk of developing Post-Traumatic Stress Disorder (PTSD) as well as other psychiatric disorders (depression, anxiety, suicidal behavior, addictions) and somatic issues that persist into adulthood. Psychological trauma can interfere with a child's psycho-affective, cognitive, and identity development, as well as with learning processes. Furthermore, trauma also affects the child's environment and family, disrupting family dynamics, relationships within the nuclear and extended family, as well as the mental health of parents and siblings. Traumatic exposure particularly impacts children and adolescents with pre-existing neurodevelopmental disorders (NDD) (e.g., Attention Deficit Hyperactivity Disorder, Autism Spectrum Disorder, specific learning disorders) and complicates their responses and engagement with their usual treatment. This is especially critical, as children with NDD are at a higher risk than the general population for maltreatment, abuse, and/or bullying .

A meta-analysis of 27 studies on PTSD in children aged 5 to 18 shows that for some exposed individuals, there is spontaneous resolution in the months following the traumatic exposure: the prevalence of PTSD in the acute phase, one month after TE, was 21%, decreasing to 15% at three months, then to 12% and 11% at six months and one year after the TE, respectively. However, given the high rates of exposure, the percentage of children at risk of developing PTSD or associated disorders remains significant. Additionally, symptoms appearing in the acute phase, such as intrusive thoughts and irritability, cause distress for the child and their family and may lead to functional impairment, interfering with optimal development.

It is currently understood that multiple individual and contextual factors before and after traumatic exposure can either facilitate or hinder the remission of acute stress symptoms and the development of PTSD and other associated disorders. A history of traumatic exposure or neurodevelopmental disorder, younger age at the time of the TE, female gender, the nature of the TE involving intentional violence by one person against another, and post-traumatic symptoms in parents are all associated with more severe post-traumatic reactions, a higher risk of developing PTSD, and a lower response to proposed treatments. Furthermore, social and family support has been shown to be a key protective factor, facilitating the management of post-traumatic reactions following a TE and preventing the onset of PTSD in children and adolescents. It is well established that parents or primary attachment figures play a crucial role in helping children build resilience in the face of adversity. A literature meta-analysis examining the role of parental behavior in the development of PTSD in children revealed that negative parenting (hostility, overprotection) is significantly associated with child PTSD. Additionally, involvement in (or reactions to) events that impact their children can be traumatic for parents themselves, which may, in turn, affect their ability to effectively support their child at a time when the child is particularly vulnerable.

There is thus a crucial need for early and effective interventions to reduce the functional impact on development and to optimize the adaptive capacities of parents and children. Detecting traumatic situations and providing care in the wake of acute traumatic exposure or upon discovery of such exposure is essential to ensure favorable post-traumatic adjustment and prevent progression to psychotraumatic syndrome and other associated disorders, in addition to alleviating acute distress and functional impact.

Contrary to the abundant literature on established PTSD therapies, which are well-documented, there is limited data on early interventions within the first forty five days following exposure to traumatic events. The investigators conducted a scoping review on this subject to identify early interventions that have been tested and validated following traumatic exposure in children and adolescents. A promising intervention that emerged from the investigators literature review is the CFTSI (Child and Family Traumatic Stress Intervention), a brief early intervention developed at the Yale Child Study Center for children aged seven to seventeen who have recently experienced a traumatic event (TE). CFTSI is a family-centered intervention lasting five to eight sessions, aiming to strengthen parental support for the child by facilitating the identification of the child's typical responses to TE, improving communication between the child and the parent, and teaching coping strategies and behavioral interventions to both parents and children to reduce acute post-traumatic reactions.

The model has been implemented with children exposed to various TEs, including sexual abuse, domestic and community violence, road accidents, animal bites, and other injuries, but not chronic, ongoing TEs, such as child maltreatment or war contexts. CFTSI can be implemented within three months following exposure to a TE. In a randomized controlled trial (RCT) comparing CFTSI to a five-session psychoeducational and non-specific psychological support model, Berkowitz et al. found that children in the CFTSI group had fewer full and partial PTSD diagnoses compared to the control group three months post-intervention. Additionally, a multicenter study without a control group assessing CFTSI's effectiveness in 1,190 families found a significant reduction in acute post-traumatic symptoms in children post-CFTSI. This same study found that symptom reduction was independent of age, gender, ethnicity, number of previous traumatic exposures, type of event, or time elapsed between the traumatic event and the start of CFTSI (e.g., after a few days or weeks).

Similarly, a multisite meta-analysis examining CFTSI's effectiveness across various centers in the United States indicated a significant improvement in post-traumatic symptoms in adult parents who participated in CFTSI with their children. This is one of the few studies that specifically evaluated the effect of early intervention after a child's exposure to a TE on parental symptoms and mental health. These results align with research establishing correlations between parental and child psychopathology, as the family environment and parental functioning systematically influence the association between traumatic exposure and its consequences for children. Additionally, involvement in events that affect their children can be traumatic for parents themselves, which may affect their ability to effectively support a child rendered vulnerable after TE exposure. Parents experiencing significant emotional distress are less able to demonstrate a sense of stability and security to the child and to support the child in their recovery. Conversely, when parents cope effectively, this can facilitate the child's adjustment post-TE by modeling effective coping skills, maintaining balance through routine and regulation, and instilling self-efficacy and relational skills. This underscores the importance of interventions aimed at strengthening parental capacities following the child's exposure to a traumatic event and providing additional support to parents significantly affected by their child's TE exposure, especially as parental ability to support their children is linked to their own level of emotional distress.

A recent study evaluating the effectiveness of CFTSI's online format showed significant reductions in child and parent PTSD symptoms before and after the intervention, even among children with chronic traumatic exposure.

The investigators have thus begun implementing CFTSI in routine practice at the Montpellier Child/Adolescent Regional Center for Psychotrauma (CRP) within the Child and Adolescent Psychological Medicine Service, following certification training with Yale University: two psychiatric nurses, three psychologists, and a child psychiatrist have already been trained. However, while Berkowitz's study was indeed an RCT evaluating CFTSI's effectiveness in preventing the onset of PTSD diagnosis in children three months post-CFTSI, no RCTs have yet been conducted, in France or elsewhere, assessing CFTSI's effectiveness in reducing acute symptoms in children and parents (thus post-CFTSI) and the persistence of these effects at three months, despite acute stress and parental symptoms remaining a significant source of suffering for children and their families.

Conducting an RCT would provide a high level of evidence for CFTSI and promote it regionally and nationally as an early intervention following traumatic exposure in children and adolescents, filling a gap in validated interventions at this level, which would alleviate children's post-traumatic stress and their parents' symptoms by enhancing parental skills. Furthermore, the investigators conducted a qualitative study with parents of adolescents aged 11 to 17 who had been exposed to a TE in the past three months to explore their experiences and perceived needs during the peri-traumatic period. The investigators' findings confirmed that parents struggled to understand their children's reactions, lacked explanations and knowledge about post-traumatic stress, expressed a sense of failure and parental inefficacy in the face of their child's suffering, hesitated on the best approach to conflicting needs, felt considerable shame and guilt, and tended to alternate between avoidant educational attitudes and coercive parenting, which strained their relationship with their child and led to conflicting dynamics. These qualitative data indicate the need to offer these parents an early, validated family intervention following their child's traumatic exposure to strengthen family support, a major protective factor.

The investigators study aims to evaluate, through a randomized controlled trial, the following objectives: (i) Effectiveness of CFTSI in reducing post-traumatic symptoms in children and adolescents aged 7 to 17 who have been exposed to traumatic events (TE) within the past three months, assessed both immediately after completion of the program and at 3 months following completion ; (ii) Impact of CFTSI on parental post-traumatic symptoms, assessed both immediately after completion of the program and at 3 months following completion ; (iii) Mediators of response to CFTSI among youth.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 7 and 17 years living in the family home;
* Having been exposed to a traumatic event (TE) in the last 3 months;
* Exhibiting at least one symptom on the Child Post-Traumatic Stress Checklist (CPC);
* Having at least one of the two parents available to participate in the intervention; and
* Having a good command of French, both orally and in writing.
* No participation in other therapeutic interventions aimed at treating traumatic stress symptoms is allowed during the inclusion period.

Exclusion Criteria:

* Parents and/or children in acute and severe emotional distress and/or in a suicidal crisis. During the recruitment interview and signing of the consent letter, the principal investigator will ensure that the volunteer participants are not in acute suicidal crisis or in severe emotional distress requiring urgent care, which would prevent them from participating in a five-session intervention (CFTSI). This emotional distress assessment will be a clinical evaluation based on the clinician's judgment.
* Child in foster care or in the process of being placed.
* Suspected maltreatment or abuse of any kind by the parents.
* Child and/or parent with a known and/or documented intellectual disability.
* Absence of consent from either of the child's parents or the child's non-agreement to participate (appropriately obtained according to the child's developmental age, taking the time to explain the procedure and intervention to the child).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Evolution of post-traumatic stress symptoms before and after the Child and Family Traumatic Stress Intervention (CFTSI) | Baseline, immediately after completion of the program, and 3 months after completion of the program.
  Assessed by the variation in total symptom scores on the Child Posttraumatic Stress Checklist (CPC), child version. This scale is validated in French, with strong psychometric properties. The original English version was designed in accordance with DSM-5 diagnostic criteria. This questionnaire assesses PTSD symptoms and their frequency in children aged 7 to 18, following a traumatic event. The minimum age of 7 years has been maintained since the original validation of the English version.
  The total score can range from 0 (no symptoms) to 84 (maximum symptoms) for symptom intensity and from 0 (no functional impact) to 24 (maximum functional impact) for functional impairment.

SECONDARY OUTCOMES:
Evolution of post-traumatic stress symptoms in children at baseline, immediately after completion of the program, and 3 months after completion of the program. | Baseline, immediately after completion of the program, and 3 months after completion of the program.
  Evaluated by the variation in the total symptom score on the Child Posttraumatic Stress Checklist (CPC), child version, compared to the pre-intervention score. This scale will be administered in our study by an evaluator blind to the randomization arm at baseline, immediately after completion of the program, and 3 months after completion of the program. This same evaluator will also be blind to the number of sessions completed and the medical history of the participants. The total score can range from 0 (no symptoms) to 84 (maximum symptoms) for symptom intensity and from 0 (no functional impact) to 24 (maximum functional impact) for functional impairment.
Evolution of post-traumatic stress symptoms in parents, at baseline, immediately after completion of the program, and 3 months after completion of the program. | Baseline, immediately after completion of the program, and 3 months after completion of the program.
  The Post-Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) consists of 20 items corresponding to the 20 Post-Traumatic Stress Disorder (PTSD) criteria detailed in the DSM-5 and includes four subscales matching the four symptom clusters: intrusion phenomena, avoidance, negative alterations in cognition and mood, and increased hyperactivity and reactivity. It has been validated in French with good psychometric properties. It is a revised version of the original PCL, which had 17 items and three subscales corresponding to the older three symptom clusters of DSM-4.
  In the PCL-5, a score of 2 or more on any item (scale: 0 to 4) is considered clinically significant. The score can range from 0 (no symptoms) to 80 (maximum symptoms).
Correlation between Child Posttraumatic Stress Checklist (CPC) total score (child version) and variables from a socio-demographic and developmental questionnaire | Baseline
  Correlation between total score on the Child Posttraumatic Stress Checklist (CPC - child version) and variables from a socio-demographic and developmental questionnaire : age, gender, socio-economic status of the parents, nature of the current traumatic event (TE).
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score and presence of a pre-existing psychiatric or neurodevelopmental disorder prior to the traumatic event (TE) | Baseline
  Association between CPC total symptom score and the presence of a pre-existing psychiatric or neurodevelopmental disorder assessed by the Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS).
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score and trauma history | Baseline
  Number of prior traumatic events (TEs) using the trauma exposure history section of the first part of the Child Posttraumatic Stress Checklist (CPC), child version. This Part 1 inquires about a broad range of TEs, including abuse and neglect, interpersonal violence, medical/unintentional injuries, and natural disasters.
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score and parental trauma exposure (LEC-5) | Baseline
  Correlation between child PTSD symptoms and parental trauma history, measured by the Life Events Checklist for DSM-5 (LEC-5).
  The LEC-5 consists of a list of 16 potentially traumatic events: for each event, the participant must indicate their level of exposure (experienced it directly, witnessed it, learned about it, or it was related to their work). It does not generate a total score but allows for the recording of traumatic events, indicating whether they have occurred or not.
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score and parental Post-Traumatic Stress Disorder (PTSD) symptoms (PCL-5) at baseline | Baseline
  Parental PTSD symptoms assessed using the PTSD Checklist for DSM-5 (PCL-5), with a score range of 0 to 80. Higher scores indicate more severe symptoms.
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score and Child and Youth Resilience Measure (CYRM-28) child version | Baseline, immediately after completion of the program, and 3 months after completion of the program.
  Resilience measured using the Child and Youth Resilience Measure (CYRM-28), child version (version for 7-10 or 11-17 years old).
  The CYRM-28 consists of 17 items measuring social, familial support, and the child/adolescent's everyday skills. Its total score ranges from 28 to 140: higher scores indicate greater resilience.
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score (child version) and data from a socio-demographic and developmental questionnaire | Baseline
  Correlation between total score on the Child Posttraumatic Stress Checklist (CPC - child version) and variables from a socio-demographic questionnaire (age, gender, socio-economic status, nature of the traumatic event).
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe Post-Traumatic Stress Disorder (PTSD) symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score and the presence of traumatic exposures prior to the current traumatic event (TE) | Baseline, immediately after completion of the program, and 3 months after completion of the program.
  The presence of one or more traumatic exposures prior to the current TE is assessed by the Traumatic Exposure History Checklist in Part 1 of the CPC, Child Version. This first part inquires about a wide range of TEs, including abuse and neglect, interpersonal violence, medical/unintentional injuries, and natural disasters.
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score and parental trauma exposure (LEC-5) | Baseline
  Correlation between child PTSD symptoms and parental trauma history, measured by the Life Events Checklist for DSM-5 (LEC-5).
  The LEC-5 consists of a list of potentially traumatic events: for each event, the participant must indicate their level of exposure (experienced it directly, witnessed it, learned about it, or it was related to their work). It does not generate a total score but allows for the recording of traumatic events, indicating whether they have occurred or not.
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score and parental Post-Traumatic Stress Disorder (PTSD) symptoms (PCL-5) | Baseline, immediately after completion of the program, and 3 months after completion of the program.
  Parental PTSD symptoms assessed using the PTSD Checklist for DSM-5 (PCL-5), with a score range of 0 to 80. Higher scores indicate more severe symptoms.
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score and parental presence during the program | Immediately after completion of the program, and 3 months after completion of the program.
  Binary variable indicating whether one or both parents were present during CFTSI sessions (yes/no).
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Correlation between Child Posttraumatic Stress Checklist (CPC) total score and time elapsed before Child and Family Traumatic Stress Intervention (CFTSI) implementation | Baseline, immediately after completion of the program, and 3 months after completion of the program.
  The delay before CFTSI implementation is the time, in days, between index trauma and the first CFTSI session.
  Child Posttraumatic Stress Checklist (CPC) total symptom score ranges from 0 to 84: higher scores indicate more severe PTSD symptoms.
Mean change in Post-Traumatic Stress Disorder (PTSD) symptoms (PTSD-Rating Index) during Child and Family Traumatic Stress Intervention (CFTSI) sessions | During the program period (weekly for 5 weeks)
  PTSD symptoms assessed using the Posttraumatic Stress Disorder-Rating Index (PTSD-RI), clinician-rated, during each CFTSI session. Score ranges from 0 to 88: higher scores indicate more severe symptoms.
  This questionnaire, administered by clinicians, is integrated into CFTSI sessions and is used in each session as a tool to enhance symptom identification and communication.
Mean change in Mood and Feelings Questionnaire (MFQ) score | During the program period (weekly for 5 weeks).
  Depressive symptoms measured using the Mood and Feelings Questionnaire. MFQ score ranges from 0 to 66 (higher scores indicate more severe depressive symptoms).
  This questionnaire, administered by clinicians, is integrated into CFTSI sessions and is used in each session as a tool to enhance symptom identification and communication.
Concordance between child- and parent-reported post-traumatic symptoms via Child Posttraumatic Stress Checklist (CPC) child and parent version | Baseline, immediately after completion of the program, and 3 months after completion of the program.
  Measured by comparing scores on the Child Posttraumatic Stress Checklist (CPC), child and parent version, and score for each symptom item. The total score can range from 0 (no symptoms) to 84 (maximum symptoms) for symptom intensity and from 0 (no functional impact) to 24 (maximum functional impact) for functional impairment.
Concordance between child- and parent-reported child's perception of social support and skills via Child and Youth Resilience Measure (CYRM) child and parent version | Baseline, immediately after completion of the program, and 3 months after completion of the program.
  Measured by comparing scores on the Child and Youth Resilience Measure (CYRM), child (7-10 or 11-17 version) and parent version.
  The CYRM score ranges from 28 to 140: higher scores indicate greater resilience.

OTHER OUTCOMES:
Sociodemograhic data | Baseline
  Additional data, beyond those that will be studied in their association with post-traumatic stress symptom scores in children on the CPC before any intervention, and with the variation in post-traumatic stress symptoms on the child version of the CPC (post-intervention and at 3 months post-intervention compared to pre-intervention, will also be collected. These include age, sibling count, nationality, and history of psychiatric/psychological follow-up.
Developmental History | Baseline
  The developmental history will collect information about the psychomotor and socio-affective development of the child or adolescent.
Session adherence : attendance to all core intervention sessions | During the program period, up to 8 weeks
  Session adherence is defined as the attendance to all five core sessions of the intervention, from start to finish, whether in the experimental or control group. If additional sessions are scheduled to address specific points, and families do not attend these extra sessions but have completed the five core sessions, adherence will be considered met (since the five core sessions were attended).

CONTACTS AND LOCATIONS:
Overall Officials: Erica EF Fongaro, Post-doc, Study Chair — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No